CLINICAL TRIAL: NCT02771730
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Orally-administered Replication-competent Adenovirus Type-4 HIV Vaccine Regimens in Combination With an AIDSVAX® B/E Boost in Healthy, HIV-uninfected Adult Participants
Brief Title: Study to Evaluate the Safety and Immunogenicity of an Oral HIV Vaccine in Healthy, HIV-uninfected Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study endpoints not met.
Sponsor: Emergent BioSolutions (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 110; 2010-0751 (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2016-05-05; First posted 2016-05-13 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteer; HIV Vaccine
MeSH Terms: interventions — AIDSVAX B-E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Vaccine A (Experimental): Receive Ad4-mgag three times at 0,2,and 6 months with a boost at 8months
  Interventions: Biological: Ad4-mgag; Biological: AIDSVAX B/E
- Vaccine B (Experimental): Receive Ad4-EnvC150 three times at 0,2,and 6 months with a boost at 8 months
  Interventions: Biological: Ad4-EnvC150; Biological: AIDSVAX B/E
- Vaccine A & B (Experimental): Receive both Ad4-mgag and Ad4-EnvC150 three times at 0,2,and 6 months with a boost at 8 months
  Interventions: Biological: Ad4-mgag; Biological: Ad4-EnvC150; Biological: AIDSVAX B/E
- Placebo (Placebo Comparator): Receive placebo three times at 0,2,and 6 months with a boost at 8 months
  Interventions: Other: Placebo Comparator; Biological: AIDSVAX B/E
- Vaccine A & B (previously received study vaccine) (Experimental): People who have previously had a study vaccine: Receive both Ad4-mgag and Ad4-EnvC150 three times at 0,2,and 6 months with a boost at 8 months
  Interventions: Biological: Ad4-mgag; Biological: Ad4-EnvC150; Biological: AIDSVAX B/E

INTERVENTIONS:
Biological: Ad4-mgag — A live replication-competent Adenovirus type-4 vector encoding a mosaic HIV Gag antigen, delivered orally by enteric-coated capsules.
  Arms: Vaccine A; Vaccine A & B; Vaccine A & B (previously received study vaccine)
Biological: Ad4-EnvC150 — A live replication-competent Adenovirus type-4 vector encoding an HIV clade C Env protein (gp150 1086.C), delivered orally by enteric-coated capsules.
  Arms: Vaccine A & B; Vaccine A & B (previously received study vaccine); Vaccine B
Other: Placebo Comparator — Oral sucrose capsules
  Arms: Placebo
Biological: AIDSVAX B/E — 300 mcg of subtype B (MN) HIV gp120 glycoprotein and 300 mcg of subtype E (A244) HIV gp120 glycoprotein adsorbed onto 600 mcg of aluminum hydroxide gel adjuvant, administered intramuscularly (IM).

SUMMARY:
The purpose of this study is to test experimental human immunodeficiency virus (HIV) vaccines that use an adenovirus vector. The adenovirus vector may help the vaccines stimulate an immune response. Researchers want to see how the immune system will respond to these vaccines as well as if they are safe to give to people. Participants cannot get HIV from these vaccines. However, researchers also want to see if the vaccine's adenovirus is contagious. Adenoviruses cause cold symptoms or mild eye infections, therefore household and intimate contacts will be asked to participate as well.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

1. Age of 18 to 49 years.
2. Access to a participating HVTN CRS and willingness to be followed for the planned duration of the study
3. Ability and willingness to provide informed consent
4. Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
5. Willing to be contacted annually after completion of scheduled clinic visits for a total of 3 years following initial study vaccination.
6. Agrees not to enroll in another study of an investigational research agent during the study period.
7. Good general health as shown by medical history, physical exam, and screening laboratory tests without clinically significant findings within the 8 weeks prior to enrollment
8. Willing to provide nasal, rectal, and cervical (for people born female) mucosal secretion samples and throat, nasal and rectal swab samples (see Appendix J)

   HIV-Related Criteria:
9. Willingness to receive HIV test results and abide by NIH guidelines for partner notification of positive HIV results
10. Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
11. Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit.

    Laboratory Inclusion Values Hemogram/CBC
12. Hemoglobin ≥ 11.0 g/dL for volunteers who were born female, ≥ 13.0 g/dL for volunteers who were born male
13. White blood cell count = 3,300 to 12,000 cells/mm3
14. Total lymphocyte count ≥ 800 cells/mm3
15. Remaining differential either within institutional normal range or with site physician approval
16. Platelets = 125,000 to 550,000/mm3 Chemistry
17. Chemistry panel: alanine aminotransferase (ALT) < 1.25 times the institutional upper limit of normal and creatinine ≤ institutional upper limits of normal.
18. Serum total bilirubin ≤ 2 mg/dL Virology
19. Negative HIV-1 and -2 blood test: Group 1 (A-D) participants must have a negative FDA-approved EIA. Group 2 participants must have a negative test result for HIV infection following the HVTN Lab Program's in-study HIV testing algorithm.
20. Negative HBsAg
21. Negative anti-Hepatitis C virus Abs (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
22. Ad4 nAb 80% inhibitory dilution < 1:100 (This criterion does not apply to participants in Group 2).

    Urine
23. Normal urine:

    * Negative urine glucose, and
    * Negative or trace urine protein, and
    * Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis with red blood cells levels within institutional normal range).

    Reproductive Status
24. Volunteers who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
25. Reproductive status: A volunteer who was born female must meet one of the following criteria:

    • Agree to consistently use effective contraception (see Appendix B) for sexual activity that could lead to pregnancy at least 21 days prior to enrollment and 28 days following the final vaccination. Effective contraception is defined as using any of the following methods: Condoms (male or female) with or without a spermicide, Diaphragm or cervical cap with spermicide, Intrauterine device (IUD), Hormonal contraception, or Any other contraceptive method approved by the HVTN 110 PSRT Successful vasectomy in the male partner (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy); or
    * Not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation; or
    * Be sexually abstinent.
26. Volunteers who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit
27. Volunteers who were born female and are 21 years of age or older must report having had (or must be willing to undergo prior to enrollment) a Pap smear test. This is not required if the volunteer has had a documented Pap smear within the previous 3 -5 years, depending on the volunteer's age and risk. The Pap smear result must be normal or ASCUS (atypical squamous cells of undetermined significance) (see USPSTF guidelines).
28. All volunteers must agree to practice abstinence (no intimate contact) for 28 days following each Ad4 vaccination.

Exclusion Criteria:

General

1. Blood products received within 120 days before first vaccination
2. Investigational research agents received within 30 days before first vaccination
3. Body mass index (BMI) ≥ 40; or BMI ≥ 35 with 2 or more of the following: age > 45, systolic blood pressure > 140 mm Hg, diastolic blood pressure > 90 mm Hg, current smoker, known hyperlipidemia
4. Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 110 study
5. Pregnant, breastfeeding, or planning pregnancy before 28 days following the final vaccination
6. Participant whose intimate contacts do not agree to enroll in the study or consent to be tested for VISP.
7. Participants who live in the same house or apartment with, have intimate contact with, or care for, any of the following:

   1. An individual under 18 years or over 65 years of age.
   2. An individual with known HIV infection
   3. An immunocompromised or immunosuppressed individual
   4. An individual with chronic respiratory disease
   5. A woman who is currently pregnant, breast feeding, or planning a pregnancy during the period of immunization.
8. Participants caring for children <18 years of age.
9. Healthcare worker who has direct contact with immunodeficient, unstable, or pediatric patients.
10. Inability to swallow 11 capsules at a clinic visit Vaccines and other Injections
11. HIV vaccine(s) received in a prior HIV vaccine trial. (Not applicable to Group 2 participants.) For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 110 PSRT will determine eligibility on a case-by-case basis.
12. Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 110 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 110 PSRT on a case-by-case basis.
13. Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 30 days after the administration of the Ad4-HIV vaccine (eg, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever).
14. Prior receipt of an Ad5-based vaccine based on self-report
15. Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (eg, tetanus, pneumococcal, Hepatitis A or B)
16. Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 30 days after first vaccination.

    Immune System
17. Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: topical corticosteroids for mild, uncomplicated dermatitis; or [4] a single course of oral/parenteral corticosteroids at doses < 2 mg/kg/day and length of therapy < 11 days with completion at least 30 days prior to enrollment.
18. Serious adverse reactions to vaccines or to vaccine components such as a history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
19. Immunoglobulin received within 60 days before first vaccination
20. History of hypogammaglobulinemia
21. Autoimmune disease, including history of Guillain-Barre syndrome
22. Immunodeficiency Clinically significant medical conditions
23. Untreated or incompletely treated syphilis infection
24. Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

    * Acute infection or a recent (within 6 months) history of chronic infection suggestive of immunodeficiency,
    * A process that would affect the immune response,
    * A process that would require medication that affects the immune response,
    * A condition requiring chronic use of medications that inhibit gastric acidity,
    * Any contraindication to injections or repeated blood draws,
    * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
    * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
    * Any condition specifically listed among the exclusion criteria below.
25. Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to receipt of live virus vaccine, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
26. Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with past or present psychoses within the past 3 years, past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
27. Current anti-tuberculosis (TB) prophylaxis or therapy
28. Chronic respiratory disorders including asthma (see below), emphysema, interstitial lung disease, pulmonary hypertension, recurrent pneumonia, or recent or ongoing respiratory tract infection. If a respiratory disorder is transient, defer immunization but do not exclude the participant.
29. Asthma exclusion criteria:

    Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report).

    Exclude a volunteer who:
    * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
    * In the past year has either of the following:

    Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids; Needed emergency care, urgent care, hospitalization, or intubation for asthma.
30. Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
31. Thyroidectomy, or thyroid disease requiring medication during the last 12 months
32. History of radiation therapy or cytotoxic/cancer therapy
33. Hypertension:

    * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤ 150 mm Hg systolic and ≤ 100 mm Hg diastolic. For these volunteers, blood pressure must be ≤ 140 mm Hg systolic and ≤ 90 mm Hg diastolic at enrollment.
    * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥ 150 mm Hg at enrollment or diastolic blood pressure ≥ 100 mm Hg at enrollment.
34. Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
35. Malignancy (Not excluded: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure. or who is unlikely to experience recurrence of malignancy during the period of the study)
36. Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
37. Asplenia: any condition resulting in the absence of a functional spleen
38. History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
39. A rectal condition that in the opinion of the clinician represents a contraindication to rectal secretion sampling, such as an active infection or inflammation of the colorectal area (such as an HSV-2 outbreak or inflamed hemorrhoids or colitis/diarrhea).
40. Any active genital tract infection such as genital sores or ulcers, penile discharge, genital warts of the penis, scrotum, labia minora, vagina, or any other symptomatic genital infection that in the opinion of the clinician represents a contraindication to sample collection.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the Ad4-mgag and Ad4-EnvC150 vaccines in humans when administered via the oral route in combination with an AIDSVAX® B/E boost. | 14 months
  To evaluate vaccine tolerability in terms of local and systemic reactogenicity signs and symptoms, laboratory measures of safety, and AEs and SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Bennett, MD, Study Director — Emergent BioSolutions
Locations (1):
- Paxvax, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No